CLINICAL TRIAL: NCT02038582
Title: An Evaluation of Strategies to Increase Testing and Linkages of HIV Positive Individuals to Care and HIV Negative Men to Male Circumcision in Sub-Saharan Africa
Brief Title: Strategies to Increase HIV Testing, Linkages to Care, and Male Circumcision in Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Connie Celum, Professor of Medicine, Epidemiology and Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 44549-A
Record Dates: First submitted 2013-12-18; First posted 2014-01-16 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: HIV
Keywords: HIV; HIV Counseling and Testing; Linkages to Care; Point of Care CD4; Point of Care Viral Load

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- POC CD4 & Clinic Accompaniment (Active Comparator): HIV positive persons not on ART at enrollment, randomized to POC CD4 testing and follow up with clinic accompaniment
  Interventions: Other: POC CD4 Testing; Behavioral: Clinic Accompaniment
- POC CD4 & Lay Counselor (Active Comparator): HIV positive persons not on ART at enrollment, randomized to POC CD4 testing and lay counselor follow up
  Interventions: Other: POC CD4 Testing; Behavioral: Lay Counselor Follow-up
- POC CD4 & Clinic Referral (Active Comparator): HIV positive persons not on ART at enrollment, randomized to POC CD4 testing and referral to clinic
  Interventions: Other: POC CD4 Testing; Behavioral: Clinic Referral
- CD4 Referral & Clinic Accompaniment (Active Comparator): HIV positive persons not on ART at enrollment, randomized to referral for CD4 testing and follow up with clinic accompaniment
  Interventions: Other: CD4 Referral; Behavioral: Clinic Accompaniment
- CD4 Referral & Lay Counselor (Active Comparator): HIV positive persons not on ART at enrollment, randomized to referral for CD4 testing and lay counselor follow up
  Interventions: Other: CD4 Referral; Behavioral: Lay Counselor Follow-up
- CD4 Referral & Clinic Referral (Active Comparator): HIV positive persons not on ART at enrollment, randomized to referral for CD4 testing and referral to clinic
  Interventions: Other: CD4 Referral; Behavioral: Clinic Referral
- Circumcision - SMS Reminder (Active Comparator): HIV negative uncircumcised males, randomized to SMS reminder for male circumcision
  Interventions: Behavioral: SMS Reminder
- Circumcision - Lay Counselor (Active Comparator): HIV negative uncircumcised males, randomized to lay counselor follow-up for male circumcision
  Interventions: Behavioral: Lay Counselor Follow-up
- Circumcision - Promotion (Active Comparator): HIV negative uncircumcised males, randomized to promotion of male circumcision at the time of HIV testing
  Interventions: Behavioral: Circumcision Promotion
- POC VL (Active Comparator): HIV positive persons on ART, randomized to POC viral load testing
  Interventions: Other: POC VL
- Laboratory based VL assay (Active Comparator): HIV positive persons on ART, randomized to laboratory based viral load testing
  Interventions: Other: Laboratory based VL assay

INTERVENTIONS:
Other: POC CD4 Testing — Point of Care CD4 testing
  Arms: POC CD4 & Clinic Accompaniment; POC CD4 & Clinic Referral; POC CD4 & Lay Counselor
Other: CD4 Referral — Referral to CD4 testing
  Arms: CD4 Referral & Clinic Accompaniment; CD4 Referral & Clinic Referral; CD4 Referral & Lay Counselor
Behavioral: Lay Counselor Follow-up — Follow-up from a lay counselor
  Arms: CD4 Referral & Lay Counselor; Circumcision - Lay Counselor; POC CD4 & Lay Counselor
Behavioral: Clinic Accompaniment — Accompaniment to the clinic by a counselor
  Arms: CD4 Referral & Clinic Accompaniment; POC CD4 & Clinic Accompaniment
Behavioral: Clinic Referral — Referral to clinic
  Arms: CD4 Referral & Clinic Referral; POC CD4 & Clinic Referral
Behavioral: SMS Reminder — SMS reminder for male circumcision
  Arms: Circumcision - SMS Reminder
Behavioral: Circumcision Promotion — Promotion of male circumcision at the time of HIV testing
  Arms: Circumcision - Promotion
Other: POC VL — POC VL testing for HIV infected persons on ART
  Arms: POC VL
Other: Laboratory based VL assay — Laboratory based viral load testing for HIV infected persons on ART
  Arms: Laboratory based VL assay

SUMMARY:
The purpose of this study is to determine efficient, scalable, evidence-based strategies to link HIV positive individuals to care and HIV negative individuals to prevention measures, such as voluntary male circumcision.

DETAILED DESCRIPTION:
New strategies for HIV testing and linkages to care are needed, since only a minority of African adults have been tested in many settings and a drop-off occurs at each step from HIV and CD4 testing, remaining in pre-ART (antiretroviral therapy) care, ART initiation, and adherence over the long term.

This study aims to determine the effects of Point-of-Care (POC) CD4 testing, POC viral load (VL) testing and several linkage strategies (lay-counselor follow-up, accompaniment to HIV clinic by lay counselor, or clinical referral) on linkage to care and treatment adherence for HIV positive persons.

This study also aims to determine the uptake of voluntary circumcision among HIV uninfected males with either promotion at point of HIV testing, Short Message Service (SMS) follow-up or lay counselor follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Reside in the study community
* Must be 16 years or older
* Able and willing to provide informed consent/assent for study procedures
* HIV negative uncircumcised men must be age 16 - 49 years and have access to secure text messaging to be randomized to strategies for male circumcision.

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2075 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Linkage to care for HIV infected persons not on treatment following a point-of care CD4 count compared to referral to clinic for CD4 testing | Up to 12 Months
  Proportion of HIV positive individuals in the POC CD4 arm who visit a clinic, obtain a staging CD4 test, initiate ART if eligible, or have a viral load <50 copies/mL within 9 months compared to those in the clinic referral arm.
Uptake of male circumcision referral among HIV-uninfected men with either promotion at point of HIV testing, SMS follow-up or lay-counselor follow-up visits | Up to 9 months
  Proportion of HIV-uninfected men who visit a male circumcision clinic or outreach venue for information about circumcision and proportion who report being circumcised by month 3 and 9 in the lay-counselor arm compared to the SMS follow-up arm, and male circumcision promotion at HIV testing arm
Linkage to care for HIV infected persons after lay counselor follow-up, accompaniment to HIV clinic by lay counselor, or clinic referral | Up to 12 months
  Proportion of HIV positive individuals not on ART at baseline who visit a clinic, obtain a staging CD4 test, initiate ART if eligible, or have a viral load <50 copies/mL within 9 months in the lay counselor follow-up arm compared to the accompaniment and clinic referral arms

SECONDARY OUTCOMES:
POC viral load testing impact on ART adherence and viral suppression compared to standard laboratory testing | Up to 12 months
  Proportion of HIV positive persons with viral load <50 copies/mL at 3 months among those who receive POC viral load testing compared to those participants who receive standard laboratory-based viral load testing.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington
Locations (2):
- Human Sciences Research Council (HSRC), Sweetwaters, KwaZulu-Natal, South Africa
- Intergrated Community Based Initivatives (ICOBI), Kabwohe, Bushenyi, Uganda

REFERENCES:
- [Derived] Barnabas RV, van Rooyen H, Tumwesigye E, Brantley J, Baeten JM, van Heerden A, Turyamureeba B, Joseph P, Krows M, Thomas KK, Schaafsma TT, Hughes JP, Celum C. Uptake of antiretroviral therapy and male circumcision after community-based HIV testing and strategies for linkage to care versus standard clinic referral: a multisite, open-label, randomised controlled trial in South Africa and Uganda. Lancet HIV. 2016 May;3(5):e212-20. doi: 10.1016/S2352-3018(16)00020-5. Epub 2016 Mar 10. PMID 27126488